CLINICAL TRIAL: NCT01389271
Title: Open-label, Uncontrolled, Prospective Long-term Observation of Inhaled Iloprost in the Treatment of Patients With Pulmonary Hypertension up to 4 Years
Brief Title: Inhaled Iloprost in the Treatment of Patients With Pulmonary Hypertension up to 4 Years
Acronym: OPTION
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 14990; VE0910TR (Other: Company internal)
Record Dates: First submitted 2011-06-27; First posted 2011-07-08 (Estimated); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary hypertension; Inhaled iloprost; Efficacy; Safety; Tolerability; Survival; NYHA class III and IV
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Iloprost

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Ventavis inhaled (Iloprost, BAYQ6256)

INTERVENTIONS:
Drug: Ventavis inhaled (Iloprost, BAYQ6256) — Since this study is an observational, inhaled iloprost dosage and frequency for each patient will be prescribed by physicians as medically required.

SUMMARY:
This is an open-label, uncontrolled, prospective long-term observation of Specific Drug in the treatment of patients with pulmonary hypertension up to 4 years. 160 patients with primary (idiopathic and familial) pulmonary hypertension (PH) or pulmonary arterial hypertension (PAH) due to scleroderma with New York Heart Association (NYHA) functional class and exercise capacity, defined as class III and IV planned to enroll. Efficacy, safety and tolerability of the drug and the survival of the patients will be observed.

ELIGIBILITY:
Inclusion Criteria:

* Patients who has pulmonary hypertension treated with inhaled iloprost older than 18 years old.
* Primary (idiopathic and familial) pulmonary hypertension (PH) with New York Heart Association (NYHA) functional class and exercise capacity, defined as class III and IV.
* Pulmonary arterial hypertension (PAH) due to scleroderma with New York Heart Association (NYHA) functional class and exercise capacity, defined as class III and IV.
* Patients who signed written informed consent.

Exclusion Criteria:

* Severe coronary heart disease or unstable angina; Myocardial infarction within the last six months; Decompensated cardiac failure if not under close medical supervision;
* Severe arrhythmias;
* Cerebrovascular events (e.g. transient ischaemic attack, stroke) within the last 3 months.
* Pulmonary hypertension due to venous occlusive disease.
* Congenital or acquired valvular defects with clinically relevant myocardial function disorders not related to pulmonary hypertension.
* Pregnancy and lactation
* Age below 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary (idiopathic and familial) pulmonary hypertension and PAH secondary to scleroderma without significant interstitial pulmonary disease classified as New York Heart Association (NYHA) functional class III and IV
Sampling Method: Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2011-02-03 (Actual); Primary Completion 2017-03-08 (Actual); Study Completion 2018-06-18 (Actual)

PRIMARY OUTCOMES:
6 Minutes walking distance (change in meters) | At month 48
Adverse events, weight, vital findings | At month 48

SECONDARY OUTCOMES:
6 Minutes walking distance (% change) | At month 48
New York Heart Association Functional Class | At month 48
Change in drug dosage or frequency, need for PAH specific drug combination, need for drug change | At month 48
Pulmonary hypertension related hospitalization | At month 48
Heart and/or lung transplantation, mortality | At month 48

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Turkey (Türkiye)